CLINICAL TRIAL: NCT07122102
Title: A Multicenter, Randomized, Open-Label, Parallel-Controlled Clinical Study Comparing the Efficacy and Safety of Cofrogliptin Versus Acarbose in Drug-Naïve Patients With Type 2 Diabetes
Acronym: CARAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK7653-503
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: cofrogliptin; acarbose; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cofrogliptin （HSK7653） (Experimental): Cofrogliptin tablets,10mg administered once every two weeks
  Interventions: Drug: Cofrogliptin
- Acarbose (Active Comparator): Acarbose tablets, 50mg administered three times daily
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Cofrogliptin — 10mg administered once every two weeks
  Arms: Cofrogliptin （HSK7653）
Drug: Acarbose — 50mg administered 3 times daily
  Arms: Acarbose

SUMMARY:
This study will compare the effect and safety of cofrogliptin (HSK7653) with acarbose among people with type 2 diabetes

DETAILED DESCRIPTION:
This study will enroll treatment-naïve patients with type 2 diabetes who meet inclusion criteria, and randomize them 1:1 to either the coglitin treatment group or the acarbose treatment group for a 12-week open-label parallel-controlled treatment period, with the coglitin group receiving 10mg coglitin tablets once every two weeks and the acarbose group receiving 50mg acarbose tablets three times daily; the primary endpoint is the change in glycated hemoglobin (HbA1c) from baseline at week 12, followed by a 1-week safety follow-up visit after treatment completion, with study conclusion upon completion of this safety visit.

ELIGIBILITY:
Inclusion Criteria:

* 1.Capable of understanding and voluntarily signing the written informed consent form.

  2.Male or female aged ≥18 years (inclusive). 3.Fulfills diagnostic criteria for type 2 diabetes mellitus. 4.Previous glycemic control managed exclusively through diet and exercise therapy, with no prior exposure to any glucose-lowering or diabetes-related medications.

  5.HbA1c at randomization: 7.0% ≤ HbA1c ≤ 9.0%. 6.Fasting plasma glucose (FPG) at randomization: FPG ≤ 11 mmol/L. 7.Body mass index (BMI) at randomization: 18 ≤ BMI ≤ 35 kg/m². 8.Agrees to maintain consistent dietary and exercise habits throughout the trial period.

Exclusion Criteria:

* 1.Known hypersensitivity to any component of the investigational product, chemically related compounds, or excipients.

  2.History of diabetic ketoacidosis, type 1 diabetes, pancreatic/β-cell transplantation, or diabetes secondary to pancreatitis/pancreatectomy.

  3.Acute coronary syndrome (STEMI/NSTEMI/unstable angina), stroke, or transient ischemic attack (TIA) within 3 months prior to informed consent.

  4.Congestive heart failure (NYHA Class III-IV). 5.Uncontrolled hypertension (systolic BP ≥180 mmHg or diastolic BP ≥110 mmHg). 6.Hepatic impairment: ALT, AST, or ALP >3×ULN at screening. 7.Severe renal impairment (eGFR <25 mL/min/1.73m²). 8.Chronic gastrointestinal disorders with significant malabsorption. 9.Conditions potentially aggravated by intestinal gas (e.g., Roemheld syndrome, severe hernia, intestinal obstruction/ulceration).

  10.Bariatric surgery or malabsorptive gastrointestinal procedures within past 2 years.

  11.Anti-obesity medications within 3 months prior to consent or weight instability at screening.

  12.Malignancy (except basal cell carcinoma) within 5 years and/or active cancer therapy.

  13.HIV infection. 14.Severe peripheral vascular disease. 15.Hematological disorders causing hemolysis/erythrocyte instability (e.g., malaria, babesiosis, hemolytic anemia).

  16.Current systemic corticosteroid use, thyroid hormone dose changes within 6 weeks, or uncontrolled endocrine disorders (excluding T2DM).

  17.Substance abuse within 3 months or chronic conditions potentially compromising compliance.

  18.Pregnancy, lactation, or unwillingness to use effective contraception (females/males).

  19.Participation in other clinical trials within 30 days prior to screening. 20.Any other condition deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | From enrollment to the end of treatment at 12 weeks
  The difference in HbA1c from the baseline

SECONDARY OUTCOMES:
FPG (Fasting plasma glucose) | From enrollment to the end of treatment at 12 weeks
  The difference in FPG from the baseline
2h-PPG (2-hour postprandial glucose) | From enrollment to the end of treatment at 12 weeks
  The difference in 2h-PPG from the baseline
Fasting C-peptide | From enrollment to the end of treatment at 12 weeks
  The difference in fasting C-peptide from the baseline
Insulin sensitivity | From enrollment to the end of treatment at 12 weeks
  The difference in insulin sensitivity from the baseline
Islet function | From enrollment to the end of treatment at 12 weeks
  The difference in Islet function from the baseline
Body weight | From enrollment to the end of treatment at 12 weeks
  The difference in body weight from the baseline
Intestinal microbial composition and functional characteristics | From enrollment to the end of treatment at 12 weeks
  The difference in intestinal microbial composition and functional characteristics from the baseline
Incidence of hypoglycemia | From enrollment to the end of safety visitation at 13 weeks
  The percentage of subjects who experienced any investigator-defined hypoglycemic adverse event
Gastrointestinal adverse events | From enrollment to the end of safety visitation at 13 weeks
  The percentage of subjects who experienced any investigator-defined gastrointestinal adverse events adverse event
Other adverse events | From enrollment to the end of safety visitation at 13 weeks
  The percentage of subjects who experienced any investigator-defined adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- He'nan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No